CLINICAL TRIAL: NCT07298863
Title: The Effect of Hydration Status on Substrate Oxidation at Rest and During Light and Moderate Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: University of Ontario Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PEP-2507
Record Dates: First submitted 2025-11-24; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hydration Status; Substrate Metabolism During Exercise
Keywords: hydration; metabolism; fluid retention

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, cross-over study (counterbalanced).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dehydrated control trial (Other): Fluid restriction during exercise and for remaining 24 hours
  Interventions: Other: Exercise Trial; Other: Experimental Trial
- Euhydrated with water (Other): Euhydrated with water to account for sweat loss and to maintain hydration over 24-hour period
  Interventions: Other: Exercise Trial; Other: Experimental Trial
- Euhydrated with electrolyte beverage (Experimental): Euhydrated with electrolyte beverage (220 mg sodium in 20 oz) to account for sweat loss and to maintain hydration over 24-hour period
  Interventions: Other: Exercise Trial; Other: Experimental Trial

INTERVENTIONS:
Other: Exercise Trial — Perform steady-state cycling exercise for approximately 1 hour at 70-80% of maximal heart rate
Other: Experimental Trial — 24h after exercise trial, following assigned 24h hydration plan, perform indirect calorimetry followed by 30 min of light cycling (~50% VO2 max) then 30 min of moderate-high cycling (~80% VO2 max).

SUMMARY:
Metabolic flexibility is the ability to properly switch between fat and carbohydrate stores to use for energy under different conditions (rest, feeding, exercise). Impairments in metabolic flexibility, also known as metabolic inflexibility, have been suggested to be an underlying cause of metabolic disease, like type 2 diabetes. Long-term low fluid intake may increase the risk of type 2 diabetes due to insulin resistance, a form of metabolic inflexibility. Further, low fluid intake has been shown to impair the ability to switch fuel preference during exercise.

While there is some evidence that low fluid intake may lead to impaired metabolic flexibility, more information is needed. Therefore, the purpose of this study is to evaluate the impact of hydration status on substrate preference at rest and during exercise at varying intensities (light and moderate). Further, we will examine whether biological sex and menstrual cycle phase impact hydration and metabolism under these same conditions.

DETAILED DESCRIPTION:
The 3-arm intervention will be completed in females during both the follicular and luteal phases for a total of 13 visits including the medical screening. In males, the 3-arm intervention will be completed once for a total of 7 visits including the medical screening.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female
* If female, subject is not pregnant (based on self-report)
* If female, subject has stopped taking birth control medication or removed long-acting reversible contraceptive >6 months at start of the study
* If female, subject has normal menstrual cycle (21-35 days)
* If female, subject is willing to track their menstrual cycle
* If female, subject has a smartphone compatible for application to track menstrual cycle (female only) and/or wearable data (females and males)
* Subject is 18-35 years of age, inclusive
* Subject body mass index (BMI) is between 18.5-25 kg/m2
* Subject is at least recreationally active (engaged in moderate-intensity, intermittent, or steady-state exercise at least 3 days per week for at least 60 min at a time)
* Subject is accustomed to cycling for at least 60 min
* Subject does not smoke (or has quit for at least 6 months)
* Subject is not taking medication that may interfere with the study (e.g., diuretics, laxatives, or weight loss drugs)
* Subject has no health conditions that would interfere with the study as indicated on the general health questionnaire (GHQ) e.g. cardiovascular, renal, or metabolic diseases
* Subject is not actively involved in weight loss intervention (dieting and/or anti-obesity medications)
* Subject is not allergic to adhesives (e.g., medical tape)
* Subject is willing to avoid alcohol consumption 24 hours prior to visit(s)
* Subject is willing to fast overnight (~8-12 hours)
* Subject is willing to refrain from vigorous exercise for 24 hours (light physical activity only)
* Subject is willing to be shaved at patch or electrode site, if necessary
* Subject is willing to eat the exact same food the day prior to each visit to the laboratory
* Able to speak, write, and read English
* Provision of written consent to participate

Exclusion Criteria:

* Subject has participated in a clinical trial within the past 30 days
* Subject has participated in any PepsiCo trial within past 36 months
* Subject has a condition or is taking medication that the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the person at undue risk
* Subject is allergic to alcohol (alcohol pre pads are used for blood draws
* If female, subject is taking birth control medication or has long-acting reversible contraceptive
* If male, subject is undergoing hormone therapy to alter testosterone levels (injections, transdermal patch, pill, etc.)
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory Exchange Ratio | Measured over the course of exercise bouts performed during the exercise and experimental trials. Compared across DEH, EUH-H2O, and EUH-Electrolyte arms.
  VCO2 / VO2 measured using indirect calorimetry measured by metabolic cart (Moxus or similar device) while exercising on cycle ergometer.

SECONDARY OUTCOMES:
Body Mass | Exercise Trial- following bladder void at baseline, post 1st and 2nd 30 min exercise sessions, and post 20 min rest Experimental Trial-following bladder void at baseline, post 10 min rest, post 1st and 2nd 30 min exercise sessions, and post 20 min rest
  kg
Plasma copeptin concentration | Exercise trial- Post 10 min rest, pre-exercise bout. Experimental trial- Post 10 min rest, pre indirect calorimetry; post 1st and 2nd 30 min exercise bout; post 20 min rest.
  pmol/L
Plasma osmolality | Exercise trial- Post 10 min rest, pre-exercise bout. Experimental trial- Post 10 min rest, pre indirect calorimetry; post 1st and 2nd 30 min exercise bout; post 20 min rest.
  mOsm/kg
Blood glucose | At medical screening to determine eligibility. Exercise trial- Post 10 min rest, pre-exercise bout. Experimental trial- Post 10 min rest, pre indirect calorimetry; post 1st and 2nd 30 min exercise bout; post 20 min rest.
  mg/dL
Blood lactate | Exercise trial- Post 10 min rest, pre-exercise bout. Experimental trial- Post 10 min rest, pre indirect calorimetry; post 1st and 2nd 30 min exercise bout; post 20 min rest.
  mmol/L
Peripheral blood mononuclear cell (PBMC) mitochondrial function | Exercise trial- Post 10 min rest, pre-exercise bout. Experimental trial- Post 10 min rest, pre indirect calorimetry; post 1st and 2nd 30 min exercise bout; post 20 min rest.
  cells/uL
Urine Specific Gravity | Exercise Trial-baseline, post 1st and 2nd 30 min exercise sessions, and post 20 min rest Experimental Trial-baseline, post resting metabolism assessment, post 1st and 2nd 30 min exercise sessions, and post 20 min rest
  au
Urine Osmolality | Exercise Trial-baseline, post 1st and 2nd 30 min exercise sessions, and post 20 min rest Experimental Trial-baseline, post resting metabolism assessment, post 1st and 2nd 30 min exercise sessions, and post 20 min rest
  mOsm/kg
Urine mass | Exercise Trial-baseline, post 1st and 2nd 30 min exercise sessions, and post 20 min rest Experimental Trial-baseline, post resting metabolism assessment, post 1st and 2nd 30 min exercise sessions, and post 20 min rest
  g
Urine Color | Exercise Trial-baseline, post 1st and 2nd 30 min exercise sessions, and post 20 min rest Experimental Trial-baseline, post resting metabolism assessment, post 1st and 2nd 30 min exercise sessions, and post 20 min rest
  Scale of 1 (most hydrated) to 7 (most dehydrated)
Fat and Carbohydrate Oxidation | Exercise Trial- resting metabolism assessed over 30 min rest period pre-exercise bout and exercise metabolism assessed over final 10 min of 1st and 2nd 30min exercise bout.
  resting metabolism measured by Cosmed Quark or similar device. Exercise metabolism measured by Moxus or similar device.
Energy Expenditure | Exercise Trial- resting metabolism assessed over 30 min rest period pre-exercise bout and exercise metabolism assessed over final 10 min of 1st and 2nd 30min exercise bout.
  kcal-resting metabolism measured by Cosmed Quark or similar device. Exercise metabolism measured by Moxus or similar device.
VO2 peak | Assessed at medical screening during a stress test with a 12-lead EKG on a cycle ergometer.
  mL/kg/min measured using indirect calorimetry (Moxus or similar device)
Fat and fat-free mass | At medical screening to determine body composition
  kg measured using BodPod
Fluid Intake | documented by subject on provided log for 24 hours prior to exercise and experimental trials. Exercise and Experimental Trial- DEH group restricted from fluid intake. EUH group fluid measured over duration of exercise bout (60 minutes).
  mL
Blood Pressure | Medical Screening to determine eligibility
  systolic/diastolic (mmHg)
Heart Rate | At medical screening to determine eligibility. Throughout entire duration of each 90-120 min exercise trial. Throughout entire duration of 120-150 min of each experimental trial.
  bpm
Standardized Exercise Intensity | Every 10 min throughout entire duration of each 60 min exercise trial to reach 70-80% of VO2 max. Every 10 min throughout entire duration of each 60 min experimental trial to reach 50-80% of VO2 max.
  W
Sweat Rate | Throughout entire duration of 60 min exercise bout of exercise trial. Throughout entire duration of 60 min exercise bout of each experimental trial.
  [Body mass loss (kg) + fluid intake (mL)]/Duration of exercise (hr)
Wearable Sensr Data | Continuous data collection over 24 hours from start of exercise trial through completion of experimental trial.
  photoplethysmogram (PPG) waveform data- optical signals obtained from photoplethysmography, which measure blood volume changes in the microvascular bed of tissue.
Rate of Perceived Exhaustion | Every 10 min throughout entire duration of each (2x) 30 min exercise bout for each exercise trial. Every 10 min throughout entire duration of each (2x) 30 min exercise bout for each experimental trial.
  Borg scale of rating of perceived exertion. Rated on a 6-20 scale from No exertion at all to maximal exertion.
Menstrual categorization | After medical screening and one month prior to first study session
  Current status (e.g., contraception, regular periods or not, etc.) tracked by physical log or an at-home menstrual cycle monitoring kit (Proov)
Adverse Events | Through study completion, an average of 3 weeks for male subjects and 8 weeks for female subjects.
  Documented changes in health and symptoms

CONTACTS AND LOCATIONS:
Locations (2):
- Gatorade Sports Science Institute, Valhalla, New York, United States
- University Of Ontario Institute Of Technology, Oshawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No